CLINICAL TRIAL: NCT06452355
Title: Clinical Trial Designed to Assess the Safety and Effectiveness of the KOKO™ Device In Treating Primary Abnormal Postpartum Uterine Bleeding ("APUB") or Hemorrhage ("PPH")
Brief Title: Safety and Effectiveness of the KOKO Device to Treat Primary Abnormal Postpartum Uterine Bleeding or Hemorrhage
Acronym: SERENE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KOKO Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOKO-PPH-001 (PSD-10212)
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Hemorrhage; Immediate Postpartum Hemorrhage; Hemorrhage, Postpartum
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Phase A is considered a Pilot Study during which 20 subjects were enrolled. Phase B will enroll up to 52 additional subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention (Experimental): The KOKO device will be administered to participants who are diagnosed with abnormal postpartum uterine bleeding or hemorrhage.
  Interventions: Device: KOKO Device

INTERVENTIONS:
Device: KOKO Device — The intrauterine drain is extended into the uterus, where low pressure vacuum is applied to the uterus through the fabric intrauterine drain. The KOKO™ device utilizes this vacuum to remove excess blood and compress the uterus reducing further blood loss.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the KOKO™ device in the control and reduction of primary abnormal postpartum uterine bleeding or hemorrhage.

DETAILED DESCRIPTION:
This IDE study is designed to evaluate the effectiveness and safety of the KOKO™ device to treat primary abnormal postpartum uterine bleeding or hemorrhage. The study is literature controlled.

ELIGIBILITY:
Inclusion Criteria:

* Adult Female, 18 years of age or older at time of consent.
* Subject is able to understand and provide informed consent to participate in the study.
* Diagnosis of abnormal postpartum uterine bleeding (500 - 999 ml for vaginal birth) or postpartum hemorrhage (1000 - 1500 ml for vaginal or Cesarean birth) with suspected atony within 24 hours after vaginal or cesarean birth.
* EBL, to be determined when investigator is ready to have the KOKO packaging opened: Vaginal birth: 500 - 1500 ml EBL or Cesarean birth: 1000 - 1500 ml EBL.
* Failed first - line intervention of uterotonics and uterine massage/bimanual uterine massage to stop bleeding. Note: Uterotonic administration may continue concomitant with and post KOKO use.

Exclusion Criteria:

* EBL >1500ml, to be determined when investigator is ready to have the KOKO packaging opened.
* Delivery at a gestational age < 34 weeks or, if multiples, uterus is judged <34 weeks size.
* For cesarean births: Cervix < 2.5 cm dilated before use of KOKO.
* Abnormal postpartum uterine bleeding or hemorrhage that the investigator determines to require more aggressive treatment, including any of the following:

  1. hysterectomy;
  2. B-lynch suture;
  3. uterine artery embolization or ligation;
  4. hypogastric ligation.
* Known uterine anomaly.
* Ongoing intrauterine pregnancy.
* Placental abnormality including any of the following:

  1. known placenta accreta;
  2. retained placenta with known risk factors for placenta accreta (e.g., history of prior uterine surgery, including prior cesarean and placenta previa);
  3. retained placenta without easy manual removal.
* Known uterine rupture.
* Unresolved uterine inversion.
* Subject has undergone intrauterine balloon therapy, uterine packing or use of other negative pressure system(s) for tamponade treatment of this episode of abnormal postpartum uterine bleeding or hemorrhage prior to use of the KOKO™ device.
* Current cervical cancer.
* Current purulent infection of vagina, cervix, uterus.
* Diagnosis of coagulopathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Conditions treated occur only in females of childbearing age (i.e., abnormal postpartum uterine bleeding or hemorrhage)
Enrollment: 72 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Rate of Participants With Cessation of Abnormal Postpartum Uterine Bleeding or Hemorrhaging | 24 Hrs
  Control of postpartum hemorrhage, defined as the avoidance of non-surgical, second line or surgical intervention to control abnormal postpartum uterine bleeding or hemorrhage after the use of the KOKO device.
Safety: Incidence, Severity and Seriousness of Device-related Adverse Events Experienced by Participants. | 6 weeks
  Incidence (i.e., rate or number of participants), severity and seriousness of device-related Adverse Events experienced by participants will be documented during the course of the study.

SECONDARY OUTCOMES:
Time to control abnormal postpartum uterine bleeding or hemorrhage | 24 Hrs
  Time from start of treatment to control of bleeding per protocol
Rate of non-surgical or surgical procedures after KOKO use | 24 Hrs
  Rate of non-surgical or surgical procedures required to control abnormal postpartum uterine bleeding or hemorrhage after KOKO use
Transfusion rate and units | 24 Hrs through discharge
  Rate of blood product transfusion required after KOKO use, and number of transfusions units administered
KOKO Device Usability | 24 Hrs
  Clinician reported assessment of KOKO device usability

CONTACTS AND LOCATIONS:
Overall Officials: Dena Goffman, MD, Principal Investigator — Columbia University; Brian Iriye, MD, Principal Investigator — Sunrise Hospital
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - Christiana Care, Newark, Delaware
  - University of Miami, Miami, Florida
  - Indiana University School of Medicine, Dept. of OBGYN, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Baptist, New Orleans, Louisiana
  - LSU Heath Sciences Center - Shreveport, Shreveport, Louisiana
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - New York-Presbyterian Medical Group Queens, Flushing, New York
  - New York-Presbyterian Hospital (NYPH)/Columbia University Irving Medical Center (CUIMC), New York, New York
  - Duke University, Durham, North Carolina
  - MetroHealth, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - UT Health Houston, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naz H, Sarwar I, Fawad A, Nisa AU. Maternal morbidity and mortality due to primary PPH--experience at Ayub Teaching Hospital Abbottabad. J Ayub Med Coll Abbottabad. 2008 Apr-Jun;20(2):59-65. PMID 19385460
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Carroli G, Cuesta C, Abalos E, Gulmezoglu AM. Epidemiology of postpartum haemorrhage: a systematic review. Best Pract Res Clin Obstet Gynaecol. 2008 Dec;22(6):999-1012. doi: 10.1016/j.bpobgyn.2008.08.004. Epub 2008 Sep 25. PMID 18819848
- [Background] McLintock C, James AH. Obstetric hemorrhage. J Thromb Haemost. 2011 Aug;9(8):1441-51. doi: 10.1111/j.1538-7836.2011.04398.x. PMID 21668737
- [Background] AbouZahr C. Global burden of maternal death and disability. Br Med Bull. 2003;67:1-11. doi: 10.1093/bmb/ldg015. PMID 14711750
- [Background] Kramer MS, Dahhou M, Vallerand D, Liston R, Joseph KS. Risk factors for postpartum hemorrhage: can we explain the recent temporal increase? J Obstet Gynaecol Can. 2011 Aug;33(8):810-819. doi: 10.1016/S1701-2163(16)34984-2. PMID 21846436
- [Background] Bateman BT, Berman MF, Riley LE, Leffert LR. The epidemiology of postpartum hemorrhage in a large, nationwide sample of deliveries. Anesth Analg. 2010 May 1;110(5):1368-73. doi: 10.1213/ANE.0b013e3181d74898. Epub 2010 Mar 17. PMID 20237047
- [Background] D'Alton ME, Rood KM, Smid MC, Simhan HN, Skupski DW, Subramaniam A, Gibson KS, Rosen T, Clark SM, Dudley D, Iqbal SN, Paglia MJ, Duzyj CM, Chien EK, Gibbins KJ, Wine KD, Bentum NAA, Kominiarek MA, Tuuli MG, Goffman D. Intrauterine Vacuum-Induced Hemorrhage-Control Device for Rapid Treatment of Postpartum Hemorrhage. Obstet Gynecol. 2020 Nov;136(5):882-891. doi: 10.1097/AOG.0000000000004138. PMID 32909970
- [Background] Suarez S, Conde-Agudelo A, Borovac-Pinheiro A, Suarez-Rebling D, Eckardt M, Theron G, Burke TF. Uterine balloon tamponade for the treatment of postpartum hemorrhage: a systematic review and meta-analysis. Am J Obstet Gynecol. 2020 Apr;222(4):293.e1-293.e52. doi: 10.1016/j.ajog.2019.11.1287. Epub 2020 Jan 6. PMID 31917139